CLINICAL TRIAL: NCT04317170
Title: The Impact of a Music Intervention on Pain and Anxiety Associated With Local Anesthesia Administration During Dermatologic Procedures
Brief Title: Music and Local Anesthesia During Dermatologic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201812098
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pain; Anxiety
Keywords: Pain; Anxiety; Lidocaine; Local anesthesia; Dermatologic procedures; Dermatology
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Participants will be played Frederic Chopin's piano sonatas through a headphone device prior to and during injection of local anesthesia.
  Interventions: Other: Music
- No Music (No Intervention): Patients will undergo their routine procedure without being played music.

INTERVENTIONS:
Other: Music — Participants will be played Frederic Chopin's piano sonatas through a headphone device prior to and during injection of local anesthesia during their routine standard of care dermatologic procedure
  Arms: Music

SUMMARY:
The goal of the study is to determine the effect of classical music on participants pain and anxiety associated with lidocaine administration during routine standard of care dermatologic procedures.

DETAILED DESCRIPTION:
The study is a randomized, unblinded, prospective, single center clinical trial. The purpose of the study is to determine the effect of a music intervention in reducing anxiety and pain from local anesthesia administration in subjects undergoing a routine, standard of care dermatologic procedure. The study population will consist of 100 adult subjects undergoing a dermatologic procedure on the head and neck. Subjects will be randomized 1:1 into either the placebo or music intervention group.

Individuals randomized into the placebo (P) group will undergo a set of standardized steps prior to local anesthesia injection. Other factors such as skin preparation technique, needle size, anesthesia temperature, use of unbuffered solution, needle angle and approximate depth of injection will remain standardized. Individuals randomized into the music intervention (MI) group will undergo the same set of standardized steps and then be played Frederic Chopin's piano sonatas through a headphone device prior to injection. After local anesthesia administration, subjects in both treatment arms will be asked to fill out a demographics, pain and anxiety questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing dermatologic procedures on the head and neck
* Ages 18-89 years old
* English speaking
* Willingness and the ability to understand and provide informed consent

Exclusion Criteria:

* Subjects who are allergic to lidocaine
* History of bleeding tendency or coagulopathy
* Pregnant or lactating
* Active skin infection in the treatment area
* Active cancer diagnosis
* Unable to understand the protocol or give informed consent
* Any other condition, in the professional opinion of the investigator, that would potentially affect response or participation in the clinical study, or would pose as an unacceptable risk to the subject

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Pain: visual analog scale (VAS) | Assessed one time immediately after dermatologic procedure is complete
  Subjects will rate the pain using the visual analog scale (VAS), which is a 10 cm line ranging from "no pain" (far left) to "extremely painful" (far right) where patients mark their pain score with a vertical line
Anxiety | Assessed one time immediately after dermatologic procedure is complete
  Subjects will rate their anxiety using the short form of the state trait anxiety inventory (STAI), which asks participants 6 questions about their anxiety levels and asks them to rank their response from 1-4.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strazar AR, Leynes PG, Lalonde DH. Minimizing the pain of local anesthesia injection. Plast Reconstr Surg. 2013 Sep;132(3):675-684. doi: 10.1097/PRS.0b013e31829ad1e2. PMID 23985640
- [Background] Vachiramon V, Sobanko JF, Rattanaumpawan P, Miller CJ. Music reduces patient anxiety during Mohs surgery: an open-label randomized controlled trial. Dermatol Surg. 2013 Feb;39(2):298-305. doi: 10.1111/dsu.12047. Epub 2013 Jan 24. PMID 23346989
- [Background] Taddio A, Ipp M, Thivakaran S, Jamal A, Parikh C, Smart S, Sovran J, Stephens D, Katz J. Survey of the prevalence of immunization non-compliance due to needle fears in children and adults. Vaccine. 2012 Jul 6;30(32):4807-12. doi: 10.1016/j.vaccine.2012.05.011. Epub 2012 May 19. PMID 22617633
- [Background] Boerner KE, Birnie KA, Chambers CT, Taddio A, McMurtry CM, Noel M, Shah V, Pillai Riddell R; HELPinKids&Adults Team. Simple Psychological Interventions for Reducing Pain From Common Needle Procedures in Adults: Systematic Review of Randomized and Quasi-Randomized Controlled Trials. Clin J Pain. 2015 Oct;31(10 Suppl):S90-8. doi: 10.1097/AJP.0000000000000270. PMID 26352921
- [Background] Kouba DJ, LoPiccolo MC, Alam M, Bordeaux JS, Cohen B, Hanke CW, Jellinek N, Maibach HI, Tanner JW, Vashi N, Gross KG, Adamson T, Begolka WS, Moyano JV. Guidelines for the use of local anesthesia in office-based dermatologic surgery. J Am Acad Dermatol. 2016 Jun;74(6):1201-19. doi: 10.1016/j.jaad.2016.01.022. Epub 2016 Mar 4. PMID 26951939
- [Background] Huron D. Is music an evolutionary adaptation? Ann N Y Acad Sci. 2001 Jun;930:43-61. doi: 10.1111/j.1749-6632.2001.tb05724.x. PMID 11458859
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Chen X, Seth RK, Rao VS, Huang JJ, Adelman RA. Effects of music therapy on intravitreal injections: a randomized clinical trial. J Ocul Pharmacol Ther. 2012 Aug;28(4):414-9. doi: 10.1089/jop.2011.0257. Epub 2012 Apr 16. PMID 22506884
- [Background] Jacobson AF. Intradermal normal saline solution, self-selected music, and insertion difficulty effects on intravenous insertion pain. Heart Lung. 1999 Mar-Apr;28(2):114-22. doi: 10.1053/hl.1999.v28.a95256. PMID 10076111